CLINICAL TRIAL: NCT00737139
Title: A Prospective, Randomized, Double-Blind Controlled Clinical Trial to Evaluate the Post-Operative Blood Loss and Transfusion Rate Following Total Joint Arthroplasty With Intra-articular Injection of Bupivacaine and Epinephrine
Brief Title: Study Comparing Peri-articular Injection of Bupivacaine With and Without Epinephrine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Prohibitively expensive and efficacy of tranexamic acid rendered topic clinically less relevant.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Craig J Delle Valle, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDV-08012802
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Osteoarthritis
Keywords: Hip; Knee; Arthroplasty; Epinephrine; Hemostasis
MeSH Terms: conditions — Osteoarthritis | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Intra-articular Injection of Marcaine/Epinephrine
  Interventions: Procedure: Peri-articular injection of marcaine/epinephrine
- 2 (Active Comparator): Intra-articular Injection of Marcaine alone
  Interventions: Procedure: Peri-articular injection of marcaine alone

INTERVENTIONS:
Procedure: Peri-articular injection of marcaine/epinephrine — 60ml of 0.5% Bupivacaine and Epinephrine 1:200,000 Inj
  Arms: 1
Procedure: Peri-articular injection of marcaine alone — 60ml of 0.5% Bupivacaine
  Arms: 2

SUMMARY:
This study involves research. The purpose of this research is to formally investigate the hemostatic efficacy of epinephrine to minimize blood loss after total joint arthroplasty. It is unclear if using intra-articular injections of epinephrine in total joint replacement is associated with a decrease in post-operative blood loss. The initial hypothesis is: the use of intra-articular injection of epinephrine is associated with decreased post-operative blood loss.

DETAILED DESCRIPTION:
Total hip and knee arthroplasties are associated with considerable blood loss, and can conservatively range from 480 ml to 1.39 liters. Current research has focused on the prevention of allogeneic blood transfusion with the pre-operative donation and use of epoetin alfa. While the pre-operative use of epoetin alpha is associated with a substantial decrease in the rate of transfusion, there still warrants investigation into the conservation of blood volume after total joint arthroplasty.

Although epinephrine has been in use as a local hemostatic agent, the use of epinephrine injection in joint replacement is limited. The mechanism of hemostasis by epinephrine is physiologic vasoconstriction. Despite the plethora of hemostatic agents available on the market today, the rationale for the use of epinephrine in this study is the medication's mechanism of action and safety. Epinephrine's alpha receptor-mediated vasoconstriction is must be balanced with vasodilation caused by its stimulation of beta-2 receptors. The relative concentration of epinephrine determines the degree of vasoconstriction versus dilation. A better understanding of the hemostatic properties and potential of intra-articular epinephrine injection will help minimize post-operative blood loss. In turn, this may decrease the number of units transfused, increase the patient's progression in physical therapy, and shorten the hospital length of stay. The goal of this prospective, randomized, double-blinded controlled clinical trial is to compare the post-operative blood loss and transfusion rate following total joint arthroplasty with intra-articular injection of marcaine and epinephrine versus the post-operative blood loss and transfusion rate following total joint arthroplasty with intra-articular injection of marcaine alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female of any race
* Ages 18-80yr
* Patients must be undergoing hip or knee arthroplasty
* Patients must be able to understand and be willing to cooperate with study procedures
* Patient must not take platelet inhibiting drugs for 10 days before surgery
* Able to provide written and verbal informed consent
* Preoperative hemoglobin above 12g/dl
* Osteoarthritis as the primary indication for knee arthroplasty, and either osteoarthritis or avascular necrosis as the indication for total hip arthroplasty

Exclusion Criteria:

* Allergy or intolerance to the study materials or medications
* Surgical intervention during the past month for the treatment of the painful joint or its underlying etiology
* History of any substance abuse or dependence within the last 6 months
* Patients who have received an investigational drug or device in the past 30 days
* Affected joint has undergone prior open surgery
* Patient received epoetin alfa 30 days before surgery
* Pre-operative autologous blood donation
* Use of platelet inhibiting drugs 10 days prior to surgery

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Record the post-operative blood volume lost in a standard, non-reinfusion drain, number of transfused units received, and calculated blood loss index during the patient's hospital course. | Daily for 6 weeks postoperatively

SECONDARY OUTCOMES:
Record of post-operative course and health maintenance to the 6 week follow-up visit. Range of motion, patient global impressions of change (PGIC) at pre-operative, immediate, 1-day, 3-day and 6-week post-operative time points. | Daily for 6 weeks post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Craig J. Della Valle, MD, Principal Investigator — Rush University Medical Center, Department of Orthopaedics
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States